CLINICAL TRIAL: NCT05198804
Title: A Phase 1/2 Dose-Escalation and Dose-Expansion Study of ZN-c3 in Combination With Niraparib and ZN-c3 Monotherapy in Subjects With Platinum-Resistant Ovarian Cancer
Brief Title: A Study of ZN-c3 and Niraparib in Subjects With Platinum-Resistant Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c3-006; GOG-3067 (Other: GOG); 2021-004161-13 (EudraCT Number)
Record Dates: First submitted 2021-12-08; First posted 2022-01-20 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer; Platinum-resistant Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Cancer
Keywords: Wee1; Wee-1
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZN-c3 and Niraparib (Experimental): ZN-c3 in combination with Niraparib
  Interventions: Drug: ZN-c3; Drug: Niraparib
- ZN-c3 (Experimental): ZN-c3 Monotherapy
  Interventions: Drug: ZN-c3

INTERVENTIONS:
Drug: ZN-c3 — ZN-c3 will be administered.
Drug: Niraparib — Niraparib will be administered.
  Arms: ZN-c3 and Niraparib

SUMMARY:
This is a Phase 1/2 study to evaluate the safety, clinical activity, pharmacokinetics (PK), and pharmacodynamics (PD) of ZN-c3 in combination with niraparib and of ZN-c3 Monotherapy in subjects with platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
This is a Phase 1/2 open-label, multicenter study to evaluate the safety, clinical activity, PK, and PD of ZN-c3 in combination with niraparib and of ZN-c3 Monotherapy in subjects with platinum-resistant ovarian cancer who have failed Poly (ADP-ribose) polymerase inhibitor (PARPi) maintenance treatment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed recurrent high grade epithelial ovarian, primary peritoneal, or fallopian tube cancer with histologic subtypes of serous, clear cell or endometroid for which there is no known or established treatment available with curative intent.
2. Subjects must have platinum-resistant disease.
3. Must have evaluable or measurable disease according to RECIST v1.1 criterion: defined as at least one lesion that can be accurately measured.
4. Adequate hematologic and organ function.
5. Ability and willingness to take oral medication.
6. Subjects must provide formalin-fixed, paraffin-embedded tumor samples available from the primary or recurrent cancer.

Key Exclusion Criteria:

1. Prior therapy directed at the malignant tumor within the last four weeks prior to Cycle 1 Day 1 (6 weeks for nitrosoureas or mitomycin C).
2. A minimum of 10 days between termination of the prior PARPi and administration of ZN-c3 and niraparib treatment is required.
3. Any investigational drug therapy <28 days.
4. Prior treatment with a WEE1 inhibitor.
5. Known hypersensitivity to any drugs similar to ZN-c3 and/or niraparib in class or its excipients.
6. Participant has any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
7. Uncontrolled hypertension (Diastolic BP > 90 mmHg or Systolic BP > 140 mmHg).
8. Myocardial impairment of any cause (e.g., cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV).
9. Significant gastrointestinal abnormalities, requirement for IV alimentation, active peptic ulcer, chronic diarrhea, or vomiting considered to be clinically significant in the judgment of the Investigator, or prior surgical procedures affecting absorption.
10. 12-lead ECG demonstrating a corrected QT interval using Fridericia's formula (QTcF) of >480 ms, except for subjects with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid.
11. History or current evidence of congenital or family history of long QT syndrome or Torsades de Pointes (TdP).
12. Taking medications with a known risk of TdP (according to current information provided at https://crediblemeds.org).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 117 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: To investigate the safety and tolerability of ZN-c3 in combination with niraparib, including identification of the MTD and RP2D | 6 months
  Incidence and severity of Dose Limiting Toxicities (DLTs) in DLT-evaluable subjects during Cycle 1
Phase 2: To investigate the antitumor activity of ZN-c3 in combination with niraparib - Progression Free Survival at 4 months | 12 months
  Stage 1 (Futility): Progression-Free Survival at 4 months (PFS@4) as defined by the revised Response Evaluation Criteria in Solid Tumors (RECIST) Guideline version 1.1
Phase 2: To investigate the antitumor activity of ZN-c3 in combination with niraparib - Objective Response Rate | 18 months
  Stage 2 (Promising Clinical Activity): Objective response rate (ORR) as defined by the revised RECIST Guideline version 1.1 and assessed by Independent Central Review (ICR)
To determine the safety and tolerability of ZN-c3 monotherapy | 12 months
  Frequency and severity of AEs and dose modifications
To investigate the antitumor activity of ZN-c3 monotherapy | 12 months
  ORR as defined by the revised RECIST Guideline version 1.1 and assessed by ICR.

SECONDARY OUTCOMES:
To further investigate the antitumor activity of ZN-c3 in combination with niraparib and ZN-c3 monotherapy | 30 months
  Duration of response (DOR) as key secondary endpoint
To further investigate the antitumor activity of ZN-c3 in combination with niraparib and ZN-c3 monotherapy | 30 months
  Clinical Benefit Rate (CBR), Progression Free Survival (PFS) (median and 4-month rate), as defined by the revised RECIST version 1.1
To further investigate the antitumor activity of ZN-c3 in combination with niraparib and ZN-c3 monotherapy | 30 months
  Objective Response Rate (ORR) based on investigator assessment
To investigate the OS of subjects receiving ZN-c3 in combination with niraparib and ZN-c3 monotherapy | 30 months
  OS (median and at 12 months)
To investigate the safety and tolerability of ZN-c3 in combination with niraparib and ZN-c3 monotherapy | 30 months
  Frequency and severity of AEs and dose modifications
To evaluate changes in Patient Reported Outcomes (PROs) and quality of life | 30 months
  Ongoing measurement of subject-reported symptomatic toxicity according to the PRO-CTCAE, and determination of change from Baseline in self-reported quality of life using EQ-5D-5L
To investigate the plasma PK of ZN-c3 and niraparib when given in combination - Maximum Plasma Concentration | 30 months
  The maximum plasma concentration (Cmax) of ZN-c3 (and its potential metabolites, as applicable) and niraparib (and their potential metabolites, as applicable) will be determined
To investigate the plasma PK of ZN-c3 and niraparib when given in combination - Area under the plasma concentration-time curve from 0 to 24h | 30 months
  Area under the plasma concentration-time curve from 0 to 24h [AUC0-24h] of ZN-c3 (and its potential metabolites, as applicable) and niraparib (and their potential metabolites, as applicable) will be determined
To investigate the plasma PK of ZN-c3 and niraparib when given in combination - Trough concentration | 30 months
  Trough concentration [Ctrough] of ZN-c3 (and its potential metabolites, as applicable) and niraparib (and their potential metabolites, as applicable) will be determined
To investigate the plasma PK of ZN-c3 and niraparib when given in combination - Time to maximum plasma concentration | 30 months
  Time to maximum plasma concentration (Tmax) of ZN-c3 (and its potential metabolites, as applicable) and niraparib (and their potential metabolites, as applicable) will be determined

OTHER OUTCOMES:
To investigate the PD and downstream effects of ZN-c3 when given in combination with niraparib - Baseline Cyclin E expression | 30 months
  Baseline Cyclin E expression in pre-dose tumor tissue
To investigate the PD and downstream effects of ZN-c3 when given in combination with niraparib - Molecular determinants of sensitivity to ZN-c3 | 30 months
  Molecular determinants of sensitivity to ZN-c3 including but not limited to Baseline DNA Damage Repair (DDR) gene mutations, deletions, copy number variations or indices of genetic instability in either tumor tissue or cell-free DNA (cfDNA)
To investigate the PD and downstream effects of ZN-c3 when given in combination with niraparib - Changes in genomic or protein biomarkers | 30 months
  Changes in genomic or protein biomarkers in peripheral blood samples

CONTACTS AND LOCATIONS:
Locations (20):
- United States (14):
  - Arizona Oncology Associates (Wilmot HOPE) - USOR, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Karmanos Cancer Institute, Detroit, Michigan
  - Spectrum Health System, Grand Rapids, Michigan
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Optimum Clinical Research Group- Women's Oncology, Albuquerque, New Mexico
  - The Blavatnik Family - Chelsea Medical Center at Mount Sinai, New York, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- France (6):
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Lyon Sud, Saint-Genis-Laval
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - EDOG - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No